CLINICAL TRIAL: NCT07230275
Title: Rectal Prolapse and Recurrent RP
Brief Title: Frailty Increase Rectal Prolapse Recurrence
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof, Zagazig University
Other Study IDs: frailty and rectal prolapse
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rectal Prolapse
Keywords: frailty
MeSH Terms: conditions — Rectal Prolapse; Frailty | interventions — phosphatidylserine receptor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic ventral rectopexy: LVMR for management of rectal prolapse
  Interventions: Procedure: LVMR for RP
- perineal stapler resection: PSR for management of RP
  Interventions: Procedure: PSR for RP

INTERVENTIONS:
Procedure: LVMR for RP — LVMR for management of RP
  Groups: laparoscopic ventral rectopexy
Procedure: PSR for RP — PSR for management of RP
  Groups: perineal stapler resection

SUMMARY:
evaluate recurrent RP in relation to frailty

ELIGIBILITY:
Inclusion Criteria:

* EPs aged ≥60 years EFTRP (Oxford prolapse grade 5)

Exclusion Criteria:

* • aged < 60 years

  * incomplete medical records,
  * concurrent colorectal procedures,
  * multi-compartmental prolapse requiring combined operations,

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients with RP
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
recurrence in relation to frailty | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tamer.A.A.M. Habeeb, Principal Investigator — Zagazig University

IPD SHARING:
Plan to Share IPD: Yes